CLINICAL TRIAL: NCT03555955
Title: A Phase 1 Trial to Evaluate the Potential Impact of Renal Impairment on the Pharmacokinetics and Safety of CPX-351 (Daunorubicin and Cytarabine) Liposome for Injection Treatment in Adult Patients With Hematologic Malignancies
Brief Title: A Trial to Evaluate the Potential Impact of Renal Impairment on the Pharmacokinetics and Safety of CPX-351
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPX351-102
Record Dates: First submitted 2018-05-14; First posted 2018-06-14 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hematologic Malignancy; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — CPX-351

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Normal renal function
  Interventions: Drug: CPX-351
- Cohort 2 (Experimental): Moderate renal impairment
  Interventions: Drug: CPX-351
- Cohort 3 (Experimental): Severe renal impairment
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — CPX-351 is administered as an intravenous (IV) infusion over approximately 90 minutes.
  Other Names: Vyxeos™
  Arms: Cohort 1
Drug: CPX-351 — CPX-351 is administered as an intravenous (IV) infusion over approximately 90 minutes.
  Other Names: Vyxeos
  Arms: Cohort 2; Cohort 3

SUMMARY:
This study evaluates the pharmacokinetics and safety of CPX-351 in patients with moderate or severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily give informed consent.
2. Male or female patients, age ≥18 years at the time of consent.
3. Diagnosis of hematologic malignancy including, but not limited to, AML, ALL, and MDS. Patients may be newly diagnosed, refractory to initial treatment, or in relapse.
4. Patients with normal renal function, or moderate or severe renal impairment as categorized by creatinine clearance (CrCl)) using the Cockcroft-Gault Formula.
5. Consent of female patients to use a medically acceptable method of contraception for at least 2 months prior to the first dose of CPX-351 and consent of female patients to use a medically acceptable method of contraception throughout the entire study period and for 6 months following the last dose of CPX-351.
6. Male patients must be willing to refrain from sperm donation for 6 months following the last dose of CPX-351and must use adequate contraception throughout the entire study period and for 6 months following the last dose of CPX-351.

Exclusion Criteria:

1. Prior treatment with CPX-351 ≤ to 1 month before the start of CPX-351 in this study.
2. Patients with active (uncontrolled, metastatic) second malignancies are excluded.
3. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent obtaining informed consent.
4. Patients with known hypersensitivity to cytarabine, daunorubicin, or liposomal products.
5. Female patients who are pregnant, nursing, or lactating.
6. Participation in another clinical trial of an investigational drug or medical device within 30 days or 5 half-lives (whichever is longer) prior to enrollment in this study.
7. Any other condition that would cause a risk to patients if they participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of CPX-351 | Blood samples will be collected during first induction on Day 1 predose, Day 5 predose, 45 and 90 minutes post infusion start, 2, 3, 4, 6, 8, 24, 48, 96, 168, and 216 hours post Day 5 infusion start.
  The key PK parameter AUCtau will be assessed

SECONDARY OUTCOMES:
PK parameter of the individual components of CPX-351, and their respective metabolites | Blood samples will be collected during first induction on Day 1 predose, Day 5 predose, 45 and 90 minutes post infusion start, 2, 3, 4, 6, 8, 24, 48, 96, 168, and 216 hours post Day 5 infusion start.
  The key PK parameter AUCtau will be assessed
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 31 months.
  TEAEs are defined as any AE starting after the initiation of the first infusion.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northside Hospital - Blood and Bone Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - New York Medical/Westchester, Valhalla, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University Health Network/Princess Margaret Cancer Center, Toronto, Ontaro

REFERENCES:
- [Derived] Solomon SR, Powell BL, Koprivnikar J, Lai C, Male H, Michaelis LC, Newell LF, Sanford D, Jenkins J, Zelaya A, Coppola S, Faderl S, Walter RB. CPX-351 Pharmacokinetics and Safety in Adults with Hematologic Malignancies and Renal Function Impairment: Phase 1 Trial. Cancers (Basel). 2024 Feb 24;16(5):915. doi: 10.3390/cancers16050915. PMID 38473278